CLINICAL TRIAL: NCT04839601
Title: RNS® System Responsive Stimulation for Adolescents With Epilepsy Study
Brief Title: RNS System RESPONSE Study
Acronym: RESPONSE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate Enrollment
Sponsor: NeuroPace (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP10014
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Epilepsy; Partial Seizure; Neurostimulator; Complications; Drug Resistant Epilepsy; Focal Epilepsy
Keywords: Adolescent; Medically refractory; Responsive neurostimulation; Focal onset seizures; RNS System
MeSH Terms: conditions — Epilepsy; Seizures; Drug Resistant Epilepsy; Epilepsies, Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Evaluation Group (stimulation ON) (Experimental): Group of participants that have an RNS System implanted and are being treated with responsive stimulation.
  Interventions: Device: RNS System

INTERVENTIONS:
Device: RNS System — The RNS System provides closed loop responsive brain stimulation. The Neurostimulator monitors the electrical activity of the brain to detect abnormal activity that could lead to a seizure. If abnormal activity is detected, the neurostimulator delivers electrical stimulation to the brain through the leads to help prevent the seizure before it occurs.

SUMMARY:
To demonstrate that the RNS System is safe and effective as an adjunctive therapy in individuals age 12 through 17 years with medically refractory partial onset epilepsy.

DETAILED DESCRIPTION:
NeuroPace is sponsoring the RESPONSE Study with the RNS System in individuals age 12 through 17 with partial (focal) onset seizures who have undergone diagnostic testing that localized no more than 2 epileptogenic foci, are refractory to two or more antiepileptic medications, and currently have frequent and disabling seizures. For the purposes of this study, disabling seizures are defined as motor partial seizures, complex partial seizures, and/or secondarily generalized seizures. The RNS System is currently approved by the FDA for use in patients 18 years and older with hard-to-treat partial-onset seizures. The same device will be used in the RESPONSE Study.

The study is a prospective open label single arm pivotal study and participants will be followed for 2 years after placement of the RNS System. The study will enroll a maximum of 200 subjects within the United States to ensure that at least 150 subjects are implanted with the RNS System.

The study design includes one interim analysis which will occur after the 75th implanted patient reaches 12 months post-implant. If the study achieves its primary safety and effectiveness endpoint goals at the interim analysis, the study will be considered successful and enrollment will be stopped.

If the interim analysis does not achieve the primary safety and effectiveness endpoint goals, the study will continue enrolling up to the maximum of 200 patients. A final analysis will be conducted after the 150th implanted patient reaches 12 months post-implant.

ELIGIBILITY:
Inclusion Criteria:

* Subject has disabling motor simple partial seizures, complex partial seizures, and/or secondarily generalized seizures. Disabling refers to seizures that are severe enough to cause injuries, or significantly impair functional ability in domains including employment, psychosocial education and mobility.
* Subject has seizures that are distinct, stereotypical events that can be reliably counted, in the opinion of the investigator, by the subject or parent/caregiver.
* Subject had an average of three or more disabling motor simple partial seizures, complex partial seizures and/or secondarily generalized seizures over the two most recent consecutive 30-day periods, with no 30-day period with less than two seizures per subject and/or parent/caregiver report.
* Subject failed treatment with a minimum of two anti-seizure medications (used in appropriate doses) with adequate monitoring of compliance and the effects of treatment, as determined by the investigator.
* Subject has undergone diagnostic testing as part of his/her standard care that has identified no more than two epileptogenic regions.
* Subject is male or a female of childbearing potential using a reliable method of contraception (hormonal, barrier method, surgical or abstention).
* Subject is age 12 or older but will be less than age 18 (has not reached 18th birthday) at the time of implantation with the RNS System.
* Subject is able to maintain an electronic diary alone or with the assistance of a competent individual.
* Subject is able to attend clinic appointments in accordance with the study schedule.
* Subject and/or parent/guardian must be willing and able to provide informed consent and assent when appropriate.
* Subject is not currently implanted with an RNS Neurostimulator or NeuroPace Leads.
* In the investigator's opinion, subject is able to tolerate a neurosurgical procedure.

Exclusion Criteria:

* Subject has been diagnosed with primarily generalized seizures.
* Subject requires procedures that are contraindicated based on current RNS System labeling.
* In the opinion of the investigator, the subject has a clinically significant or unstable medical condition (including alcohol and/or drug abuse) or a progressive central nervous system disease.
* Subject has been diagnosed with active psychosis, major depression or suicidal ideation in the preceding year. Subjects with post-ictal psychiatric symptoms need not be excluded.
* Subject is pregnant.
* Subject is participating in a therapeutic investigational drug or other device study.
* Subject is implanted with an electronic medical device that delivers electrical energy to the brain.
* Subject has been diagnosed with psychogenic or non-epileptic seizures.
* Subject has experienced unprovoked status epilepticus in the preceding year.
* Subject is taking chronic anticoagulants.

Note: For contraindications, refer to current physician labeling (manuals) for the RNS System available at the NeuroPace website (www.neuropace.com).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Short-term chronic serious adverse device effect (SADE) rate | 84-days post-implant
  The primary safety endpoint is the percent of subjects with serious device-related adverse events at 84 days (12 weeks) post-implant.
Responder rate at 12 months post implant | The primary effectiveness endpoint is the percent of subjects with a ≥ 50% reduction in seizures at 12 months post-implant compared to the pre-implant baseline.
  12 months post-implant

OTHER OUTCOMES:
Device-related Serious Adverse Event (SADE) event rate | Implant through 2 years post-implant
  The annual SADE event rate over time in subjects age 12 - 17 years implanted with the neurostimulator and/or leads during study participation will be calculated
Event rate of Serious Adverse Events (SAEs) of particular relevance | Implant through 2 years post-implant
  The annual event rate of SAEs of particular relevance (device-related or not) will be calculated over time in subjects age 12 - 17 years implanted with the neurostimulator and/or leads during study participation.
  SAEs of particular relevance include those related to:
  * infection
  * intracranial hemorrhage
  * new more disabling seizure types
  * suicidality
Affective status as measured by the Beck Depression Inventory | Implant through 2 years post-implant
  Affective status (by summary scores from the Beck Depression Inventory (BDI), either the BDI-II or Beck Youth Inventory (BYI-II), depending on age at time of the initial clinic appointment) will be described pre-implant, as well as for the post-implant months 3, 6, 9, 12 and then every four months.
Neuropsychological functioning as assessed by a sub-set of tests in the NIH Toolbox Cognition Battery | Implant through 2 years post-implant
  Neuropsychological functioning as assessed by neuropsychological testing with pediatric validated, standardized inventories to assess 3 domains that include attention, memory, and vocabulary (Flanker Inhibitory Control and Attention Test, Picture Sequence Memory Test, and Picture Vocabulary Test, respectively). These inventories are taken from the NIH Toolbox Cognition Battery and will be described by presenting summary scores for the pre-neurostimulator implant period, as well as for the annual appointments.
Percentage change in seizure frequency | Implant through 2 years post-implant
  The percentage change in seizure frequency will be summarized and reported by medians and responder rates for each 3-month interval beginning 4 months post-implant.
Quality of life as assessed by the Quality of Life in Epilepsy Inventory (QOLIE) | Implant through 2 years post-implant
  Quality of life [by summary scores from the QOLIE-AD-48 (validated for ages 12 - 17 years) or QOLIE-31-P (validated for ages 18 and older), depending on age at time of assessment] will be described pre-neurostimulator implant, as well as at yearly time points.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Morrell, MD, Principal Investigator — NeuroPace, Inc.
Locations (2):
- United States (2):
  - Spectrum Health System, Grand Rapids, Michigan
  - Westchester Medical Center, Hawthorne, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nair DR, Laxer KD, Weber PB, Murro AM, Park YD, Barkley GL, Smith BJ, Gwinn RP, Doherty MJ, Noe KH, Zimmerman RS, Bergey GK, Anderson WS, Heck C, Liu CY, Lee RW, Sadler T, Duckrow RB, Hirsch LJ, Wharen RE Jr, Tatum W, Srinivasan S, McKhann GM, Agostini MA, Alexopoulos AV, Jobst BC, Roberts DW, Salanova V, Witt TC, Cash SS, Cole AJ, Worrell GA, Lundstrom BN, Edwards JC, Halford JJ, Spencer DC, Ernst L, Skidmore CT, Sperling MR, Miller I, Geller EB, Berg MJ, Fessler AJ, Rutecki P, Goldman AM, Mizrahi EM, Gross RE, Shields DC, Schwartz TH, Labar DR, Fountain NB, Elias WJ, Olejniczak PW, Villemarette-Pittman NR, Eisenschenk S, Roper SN, Boggs JG, Courtney TA, Sun FT, Seale CG, Miller KL, Skarpaas TL, Morrell MJ; RNS System LTT Study. Nine-year prospective efficacy and safety of brain-responsive neurostimulation for focal epilepsy. Neurology. 2020 Sep 1;95(9):e1244-e1256. doi: 10.1212/WNL.0000000000010154. Epub 2020 Jul 20. PMID 32690786